CLINICAL TRIAL: NCT06185751
Title: Phase 1 Dose-Escalation and Dose-Expansion Study of the Safety and Efficacy of CS1 CAR-T (WS-CART-CS1) in Subjects With Multiple Myeloma
Brief Title: Safety and Efficacy of CS1 CAR-T (WS-CART-CS1) in Subjects With Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Paula C. & Rodger O. Riney Blood Cancer Research (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202404090
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: Chimeric Antigen Receptor; CS1
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A Dose Escalation: WS-CART-CS1 (Experimental): * Undergo apheresis procedure for WS-CART-CS1 manufacturing.
  * Anti-multiple myeloma therapy may be given after leukapheresis and up to one week prior to the start of lymphodepleting chemotherapy at the discretion of the treating physician.
  * Lymphodepleting chemotherapy on days -5, -4, and -3.
  * Three days following the last dose of lymphodepleting chemotherapy (on Day 0), WS-CART-CS1 will be infused.
  * Part A is the dose escalation portion of the study with the starting dose of 0.5 x 10^6 cells/kg of WS-CART-CS1.
  Interventions: Biological: WS-CART-CS1; Drug: Lymphodepleting chemotherapy
- Part B Dose Expansion: WS-CART-CS1 (Experimental): * Undergo apheresis procedure for WS-CART-CS1 manufacturing.
  * Anti-multiple myeloma therapy may be given after leukapheresis and up to one week prior to the start of lymphodepleting chemotherapy at the discretion of the treating physician.
  * Lymphodepleting chemotherapy on days -5, -4, and -3.
  * Three days following the last dose of lymphodepleting chemotherapy (on Day 0), WS-CART-CS1 will be infused.
  * Part B is the dose expansion portion of the study. The dose of WS-CART-CS1 will be determined in Part A of the study.
  Interventions: Biological: WS-CART-CS1; Drug: Lymphodepleting chemotherapy

INTERVENTIONS:
Biological: WS-CART-CS1 — -Subject will be hospitalized for 7 days
Drug: Lymphodepleting chemotherapy — * Cyclophosphamide 500 mg/m^2 IV on Days -5, -4, and -3
  * Fludarabine 30 mg/m^2 IV on Days -5, -4, and -3

SUMMARY:
Despite recent therapeutic advances, multiple myeloma (MM) remains an incurable disease. Although survival has improved, there are nevertheless diminishing durations of response to each subsequent line of therapy. This highlights the need for further therapeutic innovation. BCMA-targeting CAR-T cells show impressive response rates; however, their median duration of response is disappointing. The investigators propose that CS1(SLAMF7)-targeting CAR-T cells will fill a gap in the MM armamentarium.

CS1 is an attractive target in MM because it is expressed in most patients. Elotuzumab (Empliciti®), an approved anti-CS1 antibody, has proven the clinical efficacy of this target. CAR-T cells are an ideal modality to target CS1, given that two approved treatments, ide-cel (idecabtagene vicleucel, AbecmaTM) and cilta-cel (ciltacabtagene autoleucel, Carvykti™), have proven the potential for cellular immunotherapy in MM.

The investigators are testing the safety and preliminary anti-myeloma efficacy of WS-CART-CS1, a CAR-T cell therapy targeting CS1.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory multiple myeloma after 3 or more prior lines of therapy, including proteasome inhibitor (e.g. bortezomib or carfilzomib), anti-CD38 therapy (e.g. daratumumab), and anti-BCMA therapies (e.g. BCMA bispecific antibodies or BCMA CAR-T)
* Measurable disease, defined as meeting at least one of the following criteria:

  * Serum M-protein ≥ 0.5 g/dL
  * Urine M-protein ≥ 200 mg/24 h
  * Serum FLC assay: involved FLC level ≥10 mg/dL (100 mg/L) with abnormal serum FLC ratio
  * A biopsy-proven plasmacytoma
  * Bone marrow plasma cells > 30% of total bone marrow cells
* At least 18 years of age.
* ECOG performance status ≤ 1
* Adequate renal, hepatic, respiratory, and cardiovascular function, as defined below:

  * Renal function:

    * calculated creatinine clearance ≥ 50 mL/min/1.73 m2 OR
    * radioisotope glomerular filtration rate ≥ 50 mL/min/1.73 m2 OR
    * normal serum creatinine based on age/gender per institutional normal range
  * Hepatic function:

    * ALT (SGPT) ≤ 5 x ULN for age
    * Total bilirubin ≤ 2.0 x IULN (unless the patient has Grade 1 bilirubin elevation due to Gilbert's disease or a similar syndrome involving slow conjugation of bilirubin)
  * Respiratory function:

    * Minimum level of pulmonary reserve defined as oxygen saturation > 91% measured by pulse oximetry on room air
  * Cardiovascular function:

    * LVEF ≥ 45% confirmed by echocardiogram or MUGA within 28 days of screening
* The effects of CS1 CAR-T on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (at least 2 forms of contraception, including one barrier method) prior to study entry and for 12 months after CS1 CAR-T infusion. If a female subject or female partner of a male subject becomes pregnant during therapy or within 12 months following WS-CART-CS1 infusion, the investigator must be notified in order to facilitate outcome follow-up.
* Ability to understand and willingness to sign an IRB-approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Any prior systemic therapy for multiple myeloma within 14 days before planned day of leukapheresis.
* A history of other malignancy with the exception of treated non-melanomatous skin cancers and malignancies for which all treatment was completed at least 2 years before registration and the subject has no evidence of disease.
* Currently receiving any other investigational agents.
* Receipt of any cellular therapy within 8 weeks prior to the planned start of conditioning.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to CS1 CAR-T or other agents used in the study.
* History of Grade 3 CRS or ICANS with other CAR-Ts (including BCMA CAR).
* Active hepatitis B, active hepatitis C, any uncontrolled infection, or HIV infection.
* Ongoing or active infection or other serious underlying medical condition that would impair the ability to receive protocol treatment.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2040-08-31 (Estimated)

PRIMARY OUTCOMES:
Part A: Frequency and severity of treatment-emergent adverse events | From leukapheresis through 24 months after WS-CART-CS1 infusion (approximately 24 months and 1 week)
  -Graded by CTCAE v 5.0.
Part A: Frequency of dose-limiting toxicities (DLTs) | From WS-CART-CS1 infusion through 28 days
  DLTs are defined as any Grade 3 to 5 toxicity occurring within the 28 days post infusion of WS-CART-CS1 determined to be at least possibly related to WS-CART-CS1. There are some exceptions to this and there are listed in the study protocol.
Part B: Frequency and severity of treatment-emergent adverse events | From leukaphereis through 24 months after WS-CART-CS1 infusion (approximately 24 months and 1 week)
  -Graded by CTCAE v 5.0.

SECONDARY OUTCOMES:
Part A MTD and Part B: Disease-specific objective response rate (ORR) | Within 3 months of WS-CART-CS1 infusion
  -Defined as stringent complete response (sCR), plus complete response (CR), plus very good partial response (VGPR), plus partial response (PR), plus minimal response (MR) in MM within 3 months of infusion using the International Myeloma Working Group (IMWG) response criteria in MM.
Part A MTD and Part B: Minimal residual disease (MRD) negativity in the marrow | Week 12
  -Based on next-generation flow (NGF), next-generation sequencing (NGS), or both
Part A MTD and Part B: Duration of response (DoR) | -From response 24 months after WS-CART-CS1 infusion (estimated to be 24 months)
  -DoR for subjects who respond to treatment is measured from the time measurement criteria are met for response (whichever is first recorded) until the first date that relapse or progression is objectively documented.
Part A MTD and Part B: Progression-free survival (PFS) | From WS-CART-CS1 infusion through completion of follow-up (estimated to be 15 years)
  -PFS is measured from Day 0 to time of relapse, progression or death, whichever occurs first.
Part A MTD and Part B: Overall survival (OS) | From WS-CART-CS1 infusion through completion of follow-up (estimated to be 15 years)
  -OS is defined as the time from start of treatment (Day 0) to time of death.

CONTACTS AND LOCATIONS:
Overall Officials: Armin Ghobadi, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu